CLINICAL TRIAL: NCT07083609
Title: Treatment Outcomes of Direct Oral Anticoagulants in Cerebral Venous Thrombosis: A Prospective Observational Study in Vietnam
Brief Title: Treatment Outcomes of Direct Oral Anticoagulants in Cerebral Venous Thrombosis in Vietnam
Acronym: DCVT-VN25
Status: Recruiting | Type: Observational
Sponsor: Hieu Trung Dinh (Other)
Responsible Party: Sponsor-Investigator, Hieu Trung Dinh, Principal Investigator, Bach Mai Hospital
Organization: Bach Mai Hospital (Other)
Other Study IDs: DOAC-CVT-VN2025-BMH; 45-BM-HDDD (Other: Bach Mai Hospital Ethics Committee); 580-QD-DHYHN (Other: Hanoi Medical University)
Record Dates: First submitted 2025-07-07; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Venous Thrombosis
Keywords: cerebral venous thrombosis; direct oral anticoagulants; rivaroxaban; dabigatran; major bleeding; recurrent VTE; modified Rankin Scale; quality of life; prospective cohort; observational study
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Dabigatran; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DOAC Group: Adult patients with radiologically confirmed cerebral venous thrombosis who received therapeutic-dose heparin during the acute phase and subsequently initiated treatment with a direct oral anticoagulant (dabigatran or rivaroxaban) between 5 and 15 days after the start of heparin therapy
  Interventions: Drug: Dabigatran; Drug: Rivaroxaban

INTERVENTIONS:
Drug: Dabigatran — Dabigatran will be initiated between 5 and 15 days after therapeutic-dose heparin in patients with cerebral venous thrombosis (CVT), based on clinical judgment. It is administered as part of routine clinical care.
  Other Names: Pradaxa
Drug: Rivaroxaban — Rivaroxaban will be initiated between 5 and 15 days after therapeutic-dose heparin in patients with cerebral venous thrombosis (CVT), based on clinical judgment. It is administered as part of routine clinical care.
  Other Names: Xarelto

SUMMARY:
This prospective, single-arm observational cohort study aims to evaluate the real-world effectiveness and safety of direct oral anticoagulants (DOACs), specifically dabigatran or rivaroxaban, in patients with cerebral venous thrombosis (CVT). The study will be conducted at Bach Mai Hospital, a national tertiary stroke referral center in Hanoi, Vietnam.

A minimum of 69 adults with radiologically confirmed CVT will be enrolled between June 2025 and June 2027. All participants must have received therapeutic-dose heparin during the acute phase and will be transitioned to a DOAC within 5 to 15 days, per physician judgment. All treatments are part of routine care; no investigational drugs are used.

The primary outcome is a composite of major bleeding (per ISTH criteria) or recurrent venous thromboembolism (VTE) within 6 months.

Secondary outcomes include: functional outcome (Modified Rankin Scale), venous sinus recanalization, all-cause mortality, serial D-dimer levels, post-CVT chronic headache, health-related quality of life (EQ-5D-5L), clinically relevant non-major bleeding (CRNMB), symptomatic recurrent VTE, arterial thrombotic events, and early treatment discontinuation.

This study aims to generate real-world data supporting DOAC use in CVT, particularly in Asian populations where prospective evidence is limited.

DETAILED DESCRIPTION:
Cerebral venous thrombosis (CVT) is an uncommon yet potentially life-threatening cerebrovascular condition. Direct oral anticoagulants (DOACs) are increasingly adopted for CVT management, supported by recent trials (e.g., RESPECT-CVT, CHOICE-CVT, SECRET) and observational cohorts. However, prospective real-world data, especially in low- and middle-income countries like Vietnam, remain scarce.

This single-center, prospective, single-arm observational study aims to assess the safety and effectiveness of DOACs (dabigatran or rivaroxaban) in routine clinical practice among CVT patients at Bach Mai Hospital-a leading tertiary referral center in northern Vietnam.

Eligible participants are adults (≥18 years) with radiologically confirmed CVT who received therapeutic-dose heparin during the acute phase and are transitioned to a DOAC between days 5 and 15. Patients will be followed for 6 months, with scheduled evaluations of:

Clinical outcomes

D-dimer levels

Neuroimaging for venous sinus recanalization

Functional status (Modified Rankin Scale)

Health-related quality of life (EQ-5D-5L)

Safety outcomes including major bleeding, CRNMB, symptomatic recurrent VTE, arterial events, and chronic headache

Early treatment discontinuation and its causes (e.g., adverse events, patient decision)

Findings from this study will contribute important real-world evidence to guide clinical practice, especially in Asian populations underrepresented in existing prospective research.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (ICF) to participate in the study
* Age ≥ 18 years
* Confirmed diagnosis of cerebral venous thrombosis (CVT) based on clinical presentation and neuroimaging, including one or more of the following:

MRI and MRV, AND/OR CT and CTV, AND/OR MRI or CT combined with DSA

* Initiation of DOACs within 5 to 15 days after starting treatment with heparin

Exclusion Criteria:

* CVT accompanied by antiphospholipid syndrome with all three positive laboratory criteria: lupus anticoagulant, anticardiolipin antibodies, and anti-β2-glycoprotein antibodies
* CVT in pregnant patients requiring continuous anticoagulation throughout pregnancy
* CVT with coexisting bleeding disorders, including immune thrombocytopenia with platelet count <100,000/mL, hemophilia A or B, von Willebrand disease, or a history of prolonged bleeding after surgery or invasive procedures
* CVT in patients with mechanical heart valves, atrial fibrillation, and moderate to severe mitral stenosis
* CVT in patients with a glomerular filtration rate (GFR) <15 mL/min
* CVT with severe hepatic impairment
* Patients already receiving anticoagulation therapy for another underlying condition at the time of CVT diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) with radiologically confirmed cerebral venous thrombosis (CVT) who received therapeutic-dose heparin during the acute phase and are subsequently treated with a direct oral anticoagulant. All participants will be recruited from Bach Mai Hospital, the national referral center in Vietnam that receives the majority of CVT cases in the northern region.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Composite of major bleeding or recurrent venous thromboembolism | Within 6 months after CVT diagnosis
  A composite endpoint including: (1) the occurrence of VTE, defined as recurrent CVT, deep vein thrombosis of any limb, pulmonary embolism, or thrombosis involving the splanchnic, jugular, caval, renal, or catheter-related veins; and (2) major bleeding events, defined according to the criteria established by the International Society on Thrombosis and Haemostasis (ISTH)

SECONDARY OUTCOMES:
Mortality Rate | At 6 months after CVT diagnosis
  All-cause mortality
Functional outcome | At 3 and 6 months after after CVT diagnosis
  Proportion of patients with good functional outcome, defined as a score of 0-1 on the Modified Rankin Scale (mRS). The Modified Rankin Scale ranges from 0 to 6, where 0 indicates no symptoms and 6 indicates death. Lower scores reflect better functional recovery.
Number of participants with major bleeding events | At 3 and 6 months after CVT diagnosis
  Number of major bleeding events, defined according to the criteria established by the International Society on Thrombosis and Haemostasis (ISTH).
Number of participants with clinically relevant non-major bleeding (CRNMB) events | At 3 and 6 months after CVT diagnosis
  Number of CRNMB events, defined according to the criteria established by the International Society on Thrombosis and Haemostasis (ISTH)
Number of participants with symptomatic recurrent venous thromboembolism (VTE) | At 3 and 6 months after CVT diagnosis
  Number of participants who experience symptomatic recurrent venous thromboembolism (VTE), including cerebral venous thrombosis, deep vein thrombosis, pulmonary embolism, or splanchnic thrombosis.
Number of participants who discontinued anticoagulant therapy early | At 6 months after CVT diagnosis
  Number of participants who discontinued DOAC therapy before the duration recommended by their treating physician, and documented reasons for discontinuation (e.g., adverse events, patient decision, or clinical judgment). Reasons will be collected from clinical records and follow-up interviews.
Number of participants with arterial thrombotic events | At 6 months after CVT diagnosis
  Number of participants who experience arterial thrombotic events, including ischemic stroke, myocardial infarction, or other objectively confirmed arterial thromboses. Events will be confirmed by clinical assessment and/or imaging as appropriate.
Health-related quality of life (EQ-5D-5L utility index score) | At 3 and 6 months after CVT diagnosis
  Health-related quality of life will be assessed using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument. This tool evaluates five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity.
  A utility index score will be calculated using the Vietnamese EQ-5D-5L value set, ranging from -0.511 to 1.000, where:
  1.000 indicates perfect health,
  0.000 corresponds to death,
  scores below 0 indicate health states considered worse than death by the general Vietnamese population.
Serial D-dimer measurements after CVT | At 3 and 6 months after CVT diagnosis
  Plasma D-dimer levels will be measured at 3 and 6 months using a standardized quantitative assay. Values will be reported in ng/mL and interpreted in the context of post-CVT coagulation activity.
Venous recanalization | At 6 months after CVT diagnosis
  Degree of venous sinus recanalization assessed on follow-up neuroimaging (MRI/MRV or CT/CTV) at 6 months. Recanalization will be categorized as complete, partial, or absent, based on standardized radiological criteria
Frequency of chronic headache after CVT | At 6 months after CVT diagnosis
  Presence and frequency of persistent or recurrent headache fulfilling the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria for chronic post-CVT headache. Assessment will be based on patient-reported symptoms and clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ton D. Mai, Study Chair — Hanoi Medical University
Locations (1):
- Bach Mai Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the single-center design, limited sample size, and institutional policies regarding patient confidentiality

REFERENCES:
- [Background] Yang M, Rendas-Baum R, Varon SF, Kosinski M. Validation of the Headache Impact Test (HIT-6) across episodic and chronic migraine. Cephalalgia. 2011 Feb;31(3):357-67. doi: 10.1177/0333102410379890. Epub 2010 Sep 6. PMID 20819842
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Aguiar de Sousa D, Lucas Neto L, Arauz A, Sousa AL, Gabriel D, Correia M, Gil-Gouveia R, Penas S, Carvalho Dias M, Correia MA, Carvalho M, Canhao P, Ferro JM. Early Recanalization in Patients With Cerebral Venous Thrombosis Treated With Anticoagulation. Stroke. 2020 Apr;51(4):1174-1181. doi: 10.1161/STROKEAHA.119.028532. Epub 2020 Mar 2. PMID 32114929
- [Background] Mai VQ, Sun S, Minh HV, Luo N, Giang KB, Lindholm L, Sahlen KG. An EQ-5D-5L Value Set for Vietnam. Qual Life Res. 2020 Jul;29(7):1923-1933. doi: 10.1007/s11136-020-02469-7. Epub 2020 Mar 27. PMID 32221805
- [Background] Kaatz S, Ahmad D, Spyropoulos AC, Schulman S; Subcommittee on Control of Anticoagulation. Definition of clinically relevant non-major bleeding in studies of anticoagulants in atrial fibrillation and venous thromboembolic disease in non-surgical patients: communication from the SSC of the ISTH. J Thromb Haemost. 2015 Nov;13(11):2119-26. doi: 10.1111/jth.13140. No abstract available. PMID 26764429
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Field TS, Lindsay MP, Wein T, Debicki DB, Gorman J, Heran MKS, Levin LA, Lund R, Moharir M, Peeling L, Perera KS, Siegal D, Verreault S, Foley N, Martin C, Smith EE, Mountain A, Mandzia J; Canadian Stroke Best Practice Recommendations Advisory Committee, in collaboration with the Canadian Stroke Consortium. Canadian Stroke Best Practice Recommendations, 7th Edition: Cerebral Venous Thrombosis, 2024. Can J Neurol Sci. 2024 Jun 3:1-17. doi: 10.1017/cjn.2024.269. Online ahead of print. PMID 38826076
- [Background] Ulivi L, Squitieri M, Cohen H, Cowley P, Werring DJ. Cerebral venous thrombosis: a practical guide. Pract Neurol. 2020 Oct;20(5):356-367. doi: 10.1136/practneurol-2019-002415. PMID 32958591
- [Background] Saposnik G, Bushnell C, Coutinho JM, Field TS, Furie KL, Galadanci N, Kam W, Kirkham FC, McNair ND, Singhal AB, Thijs V, Yang VXD; American Heart Association Stroke Council; Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Cardiovascular and Stroke Nursing; and Council on Hypertension. Diagnosis and Management of Cerebral Venous Thrombosis: A Scientific Statement From the American Heart Association. Stroke. 2024 Mar;55(3):e77-e90. doi: 10.1161/STR.0000000000000456. Epub 2024 Jan 29. PMID 38284265
- [Background] van de Munckhof A, van Kammen MS, Tatlisumak T, Krzywicka K, Aaron S, Antochi F, Arauz A, Barboza MA, Conforto AB, Contreras DG, Heldner MR, Hernandez-Perez M, Hiltunen S, Ji X, Kam W, Kleinig TJ, Kristoffersen ES, Leker RR, Lemmens R, Poli S, Wasay M, Wu T, Yesilot N, Chen J, Cotelli MS, Demeestere J, Duan J, Ergin N, Freitas TE, Gomes A, den Hertog HM, Lindgren E, Martinez-Majander N, Metanis I, Miraclin A, Rani LJ, Reddy YM, Saleem S, Scutelnic A, Shanmugasundaram S, van den Wijngaard IR, Gencdal IY, van Eekelen R, Vellema J, Arnold M, Neto L, Middeldorp S, de Sousa DA, Jood K, Putaala J, Ferro JM, Coutinho JM; DOAC-CVT investigators. Direct oral anticoagulants versus vitamin K antagonists for cerebral venous thrombosis (DOAC-CVT): an international, prospective, observational cohort study. Lancet Neurol. 2025 Mar;24(3):199-207. doi: 10.1016/S1474-4422(24)00519-2. PMID 39986309
- [Background] Yaghi S, Shu L, Bakradze E, Salehi Omran S, Giles JA, Amar JY, Henninger N, Elnazeir M, Liberman AL, Moncrieffe K, Lu J, Sharma R, Cheng Y, Zubair AS, Simpkins AN, Li GT, Kung JC, Perez D, Heldner M, Scutelnic A, Seiffge D, Siepen B, Rothstein A, Khazaal O, Do D, Kasab SA, Rahman LA, Mistry EA, Kerrigan D, Lafever H, Nguyen TN, Klein P, Aparicio H, Frontera J, Kuohn L, Agarwal S, Stretz C, Kala N, El Jamal S, Chang A, Cutting S, Xiao H, de Havenon A, Muddasani V, Wu T, Wilson D, Nouh A, Asad SD, Qureshi A, Moore J, Khatri P, Aziz Y, Casteigne B, Khan M, Cheng Y, Mac Grory B, Weiss M, Ryan D, Vedovati MC, Paciaroni M, Siegler JE, Kamen S, Yu S, Leon Guerrero CR, Atallah E, De Marchis GM, Brehm A, Dittrich T, Psychogios M, Alvarado-Dyer R, Kass-Hout T, Prabhakaran S, Honda T, Liebeskind DS, Furie K. Direct Oral Anticoagulants Versus Warfarin in the Treatment of Cerebral Venous Thrombosis (ACTION-CVT): A Multicenter International Study. Stroke. 2022 Mar;53(3):728-738. doi: 10.1161/STROKEAHA.121.037541. Epub 2022 Feb 10. PMID 35143325
- [Background] Field TS, Dizonno V, Almekhlafi MA, Bala F, Alhabli I, Wong H, Norena M, Villaluna MK, King-Azote P, Ratnaweera N, Mancini S, Van Gaal SC, Wilson LK, Graham BR, Sposato LA, Blacquiere D, Dewar BM, Boulos MI, Buck BH, Odier C, Perera KS, Pikula A, Tkach A, Medvedev G, Canfield C, Mortenson WB, Nadeau JO, Alshimemeri S, Benavente OR, Demchuk AM, Dowlatshahi D, Lanthier S, Lee AYY, Mandzia J, Suryanarayan D, Weitz JI, Hill MD; SECRET Investigators. Study of Rivaroxaban for Cerebral Venous Thrombosis: A Randomized Controlled Feasibility Trial Comparing Anticoagulation With Rivaroxaban to Standard-of-Care in Symptomatic Cerebral Venous Thrombosis. Stroke. 2023 Nov;54(11):2724-2736. doi: 10.1161/STROKEAHA.123.044113. Epub 2023 Sep 7. PMID 37675613
- [Background] Ma H, Gu Y, Bian T, Song H, Liu Z, Ji X, Duan J. Dabigatran etexilate versus warfarin in cerebral venous thrombosis in Chinese patients (CHOICE-CVT): An open-label, randomized controlled trial. Int J Stroke. 2024 Jul;19(6):635-644. doi: 10.1177/17474930241234749. Epub 2024 Feb 26. PMID 38353219
- [Background] Ferro JM, Coutinho JM, Dentali F, Kobayashi A, Alasheev A, Canhao P, Karpov D, Nagel S, Posthuma L, Roriz JM, Caria J, Frassdorf M, Huisman H, Reilly P, Diener HC; RE-SPECT CVT Study Group. Safety and Efficacy of Dabigatran Etexilate vs Dose-Adjusted Warfarin in Patients With Cerebral Venous Thrombosis: A Randomized Clinical Trial. JAMA Neurol. 2019 Dec 1;76(12):1457-1465. doi: 10.1001/jamaneurol.2019.2764. PMID 31479105
- [Background] Saposnik G, Barinagarrementeria F, Brown RD Jr, Bushnell CD, Cucchiara B, Cushman M, deVeber G, Ferro JM, Tsai FY; American Heart Association Stroke Council and the Council on Epidemiology and Prevention. Diagnosis and management of cerebral venous thrombosis: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2011 Apr;42(4):1158-92. doi: 10.1161/STR.0b013e31820a8364. Epub 2011 Feb 3. PMID 21293023
- [Background] Alet M, Ciardi C, Aleman A, Bandeo L, Bonardo P, Cea C, Cirio J, Cossio J, Cuculic M, Esnaola MM, Garcia-Perez F, Giner F, Gomez-Schneider M, Isaac C, Lepera S, Martinez C, Martinez-Lorenzin R, Montes M, Orzuza G, Persi G, Povedano G, Pujol-Lereis V, Quiroga-Narvaez J, Romano M, Sabio R, Viglione J, Zurru MC, Saposnik G; Argentinian Stroke and Cerebrovascular Diseases Study Group - Argentine Neurological Society. Cerebral venous thrombosis in Argentina: clinical presentation, predisposing factors, outcomes and literature review. J Stroke Cerebrovasc Dis. 2020 Oct;29(10):105145. doi: 10.1016/j.jstrokecerebrovasdis.2020.105145. Epub 2020 Jul 28. PMID 32912503
- [Background] Bousser MG, Ferro JM. Cerebral venous thrombosis: an update. Lancet Neurol. 2007 Feb;6(2):162-70. doi: 10.1016/S1474-4422(07)70029-7. PMID 17239803

DOCUMENTS (1):
  • Study Protocol (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT07083609/Prot_000.pdf